CLINICAL TRIAL: NCT03597854
Title: Renal Outcome of Acute Kidney Disease in Critically Ill Patients: A Prospective Observational Study
Brief Title: Renal Outcome of Acute Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Mohan Gurjar, Principal Investigator, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2017-234-DM-EXP
Record Dates: First submitted 2018-06-26; First posted 2018-07-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Acute Kidney Disease
Keywords: Acute kidney disease; critically ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Both, acute kidney injury (AKI) and chronic kidney disease (CKD) considered as a continuum of the disease process. The renal recovery after AKI is currently assessed by measuring serum creatinine, which has its limitations including change in muscle mass, volume distribution in critically ill patients. Also, despite complete return of serum creatinine after AKI, these patients remain at increased risk for developing CKD, which suggest that there may be persistent subclinical damage to the kidney. The new term acute kidney disease (AKD) has been proposed to define the renal disease after AKI. Recently (2017), Acute Disease Quality Initiative (ADQI) 16 workgroup published a consensus document on AKD and renal recovery, which provide definition as well as research recommendation for AKD. The consensus report of the ADQI 16 workgroup (2017) recommended that there is need for studies to describe the epidemiology, clinical course, natural history of patients having AKD; and also determine optimal methods to assess functional recovery and identify novel biomarker(s), functional tests, and imaging approach which can reveal ongoing injury and repair in these patients. This is an observational study to describe epidemiology, clinical course and recovery from AKD at 90 days in critically ill patients.

DETAILED DESCRIPTION:
Introduction and Background:

There are available definitions for acute kidney injury (AKI) and chronic kidney disease (CKD), which are being used routinely in research and clinical practice. The AKI is defined as an abrupt decrease in kidney function occurring over 7 days or less, as per KDIGO (kidney disease improving global outcome) guideline. The CKD is defined as persistence of kidney disease for a period of more than 90 days.

Both, AKI and CKD considered as a continuum of the disease process. The renal recovery after AKI is currently assessed by measuring serum creatinine, which has its limitations including change in muscle mass, volume distribution in critically ill patients. Also, despite complete return of serum creatinine after AKI, these patients remain at increased risk for developing CKD, which suggest that there may be persistent subclinical damage to the kidney. The new term acute kidney disease (AKD) has been proposed to define the renal disease after AKI. Recently (2017), Acute Disease Quality Initiative (ADQI) 16 workgroup published a consensus document on AKD and renal recovery, which provide definition as well as research recommendation for AKD.

Rationale of the study supported by cited literature:

The consensus report of the ADQI 16 workgroup (2017) recommended that there is need for studies to describe the epidemiology, clinical course, natural history of patients having AKD; and also determine optimal methods to assess functional recovery and identify novel biomarker(s), functional tests, and imaging approach which can reveal ongoing injury and repair in these patients.

The relevance and expected outcome of the proposed study:

This is an observational study to describe epidemiology, clinical course and recovery from AKD at 90 days in critically ill patients.

Preliminary work done so far:

There is no systematic study so far in critically ill patients, as AKD is defined recently.

Definition of AKD:

Acute kidney disease (AKD): Acute or subacute damage and/or loss of kidney function for a duration of between 7 and 90 days after exposure to an AKI initiating event. Outcome of AKD include recovery, recurrence of AKI, progression of AKD and/or death. Stages (1, 2 and 3) of AKD are defined same as for AKIN criteria.

Specific objectives:

• To study acute kidney disease severity outcome by measuring serum creatinine and other biomarkers (NGAL, KIM-1 and Cystatin C) at 90 days.

Work plan methodology:

This is a prospective observational study to know the disease process of AKD. Patients will be included from the ICU of Department of Critical Care Medicine and Department of Nephrology. All adult critically ill patients will be consider for inclusion in this study, who had AKD (at 7 days after exposure to an AKI initiating event) because of various etiologies during his/ her current illness. After getting written informed consent from the patient or close relatives to participate in this study, patients will be included in this study. There will be no intervention in this study. Patients will be followed up in our ICU follow-up clinic and/ or nephrology OPD at 90 days of event of acute kidney injury and various biomarkers and imaging parameters will be assessed.

Sample size:

This is an observational study, where all eligible patients will be considered for possible inclusion over 15 month duration.

Consent:

Informed written consent will be obtained from all patients or close relatives for inclusion in the study.

Sample collection:

At baseline (D7, when defined as AKD), at ICU discharge, and at 90 days (D90): 3 ml blood and 3 ml urine will be collected.

Data collection:

Demographic and clinical characteristics of all ICU patients who fulfill inclusion criteria will be collected along with relevant laboratory tests done during patient management, as per treating team. ICU prognostication scores, i.e., Acute Physiologic and Chronic Health Evaluation (APACHE) II score and Sequential Organ Dysfunction Assessment (SOFA) score will also be recorded. Episodes of recurrence of AKI will be recorded. Risk factors of acute kidney injury like presence of circulatory shock, chronic diseases (heart, lung, liver), diabetes mellitus, nephrotoxic drugs, radio contrast agents will also be noted. .

Intervention:

None

Outcome:

To study the renal outcome of AKD (among survivors) at 90 days, by measuring serum creatinine, urine routine, albuminuria, serum and urine biomarkers (NGAL, Cystatin C and KIM-1), need of renal replacement therapy and renal ultrasound.

Laboratory methods:

Samples will be analysed for plasma creatinine, urinary albumin, plasma and urine biomarkers (NGAL cystatin C, and KIM-1) at baseline (D7), at ICU discharge and at 90 days (D90). Biomarker, Neutrophil Gelatinase-Associated Lipocalin (NGAL), Cystatin C and Kidney Injury Molecule-1 in plasma will be analysed by commercially available ELISA kits (RnD) as per manufacturer instructions. Renal ultrasonography will be done at baseline (D7) and at 90 days (D90).

Statistical analysis:

Descriptive analysis will be done and data will be presented as mean or median.

Duration of the study:

15 months

ELIGIBILITY:
Inclusion Criteria:

* All ICU patients who are ≥18 years and had AKD

Exclusion Criteria:

* Age <18 years
* Not known AKI initiating event day
* Any known renal disease (like CKD, nephritic or nephrotic syndrome)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult ICU patients who had AKD (at 7 days after exposure to an AKI initiating event) will be considered for inclusion.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
To know renal outcome of acute kidney disease (AKD) among ICU survivors at 90 days after exposure to an acute kidney injury initiating event. | 90 days after exposure to an acute kidney injury initiating event.
  To study the renal outcome of AKD (among survivors) at 90 days, by measuring serum creatinine.

SECONDARY OUTCOMES:
Incidence of acute kidney disease (AKD) among ICU patients | 15 months
  Percentage of ICU patients who had AKD

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjar, MD, PDCC, Principal Investigator — SGPGIMS
Locations (1):
- Department of Critical Care Medicine, SGPGIMS, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chawla LS, Bellomo R, Bihorac A, Goldstein SL, Siew ED, Bagshaw SM, Bittleman D, Cruz D, Endre Z, Fitzgerald RL, Forni L, Kane-Gill SL, Hoste E, Koyner J, Liu KD, Macedo E, Mehta R, Murray P, Nadim M, Ostermann M, Palevsky PM, Pannu N, Rosner M, Wald R, Zarbock A, Ronco C, Kellum JA; Acute Disease Quality Initiative Workgroup 16.. Acute kidney disease and renal recovery: consensus report of the Acute Disease Quality Initiative (ADQI) 16 Workgroup. Nat Rev Nephrol. 2017 Apr;13(4):241-257. doi: 10.1038/nrneph.2017.2. Epub 2017 Feb 27. PMID 28239173